CLINICAL TRIAL: NCT02854345
Title: Preliminary Study Concerning the Validity of Parathyroid Exploration on a Discovery NM 530c CZT Camera
Brief Title: Preliminary Study Concerning the Validity of Parathyroid Exploration on a CZT Camera
Acronym: PARAT-CZT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2013/212
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Hyperparathyroidism
Keywords: CZT camera; pinhole
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tomoscintigraphic parathyroid imaging on a CZT camera (Experimental): Tomoscintigraphic parathyroid imaging on a CZT camera
  Interventions: Device: Tomoscintigraphic parathyroid imaging on a CZT camera

INTERVENTIONS:
Device: Tomoscintigraphic parathyroid imaging on a CZT camera

SUMMARY:
The goal of this study is to assess the performance of parathyroid imaging on a cardiac-dedicated CZT camera, compared to planar pinhole imaging, in patients referred for primary hyperparathyroidism.

DETAILED DESCRIPTION:
The goal is to determine if parathyroid tomoscintigraphy on a CZT camera can provide at least equivalent diagnostic performance, compared with planar pinhole imaging.

ELIGIBILITY:
Inclusion Criteria:

* suffering from sporadic primary hyperparathyroidism
* referred to the Nuclear Medicine Dept for a pre-operative scintigraphy of the parathyroid glands
* who have given their written consent
* who benefit from the French Government Medical Insurance

Exclusion Criteria:

* pregnant women
* ages < 18 or > 80 years
* hyperparathyroidism recidive after a first surgery
* secondary or tertiary hyperparathyroidism
* Multiple endocrine Neoplasia (MEN) type I context or familial history of hyperparathyroidism
* absence of written consent
* non-beneficiary of the French Government Medical Insurance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Comparison of pathologic parathyroid detection performances between planar pinhole on Anger camera and tomoscintigraphy on CZT camera, gold standard being the pathological results after surgery | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Constantin Ungureanu, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No